CLINICAL TRIAL: NCT00104091
Title: A Multicenter Phase II Study of TP-38 in Those Patients With Glioblastoma Multiforme Who Have Recurred or Progressed After Previous Resection and Radiation Therapy and Are Scheduled for Gross Total Resection
Brief Title: Safety and Efficacy Study to Treat Recurrent Grade 4 Malignant Brain Tumors
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Teva Branded Pharmaceutical Products R&D, Inc. (Industry)
Responsible Party: Rivka Kreitman, Ph.D., Vice President, Innovative Research and Development, Teva Neuroscience
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IXR-202-22-188
Record Dates: First submitted 2005-02-22; First posted 2005-02-23 (Estimated); Last update posted 2011-05-23 (Estimated); Status verified 2011-05

CONDITIONS: Glioblastoma Multiforme
Keywords: Gross Total Resection; Convection Enhanced Delivery; Recurrent Glioblastoma Multiforme
MeSH Terms: conditions — Glioblastoma | interventions — transforming growth factor(alpha)-Pseudomonas aeruginosa exotoxin (38)

ARMS (1):
- 1 (Experimental): 40 mL of TP-38 at a 100 nanograms/mL concentration
  Interventions: Drug: TP-38

INTERVENTIONS:
Drug: TP-38 — TP-38 is a recombinant chimeric protein composed of the epidermal growth factor (EGFR) binding ligand (TGF-α)and a genetically engineered form of the Pseudomonas exotoxin, PE-38.

SUMMARY:
Immunotoxin therapy may be effective in treating malignant glioma. Immunotoxins can locate tumor cells and kill them without harming normal cells.

ELIGIBILITY:
Inclusion Criteria:

The patients must fulfill all the following criteria:

* Previous histologically-confirmed diagnosis of primary GBM (glioblastoma multiforme, glioma grade 4 at time of first diagnosis).
* Histologically-confirmed and MRI diagnosed recurrent or progressive GBM after previous resection (surgical or biopsy) and radiation therapy.
* Medically capable of undergoing the planned surgical gross total resection and the catheter placement.
* Age ≥ 18.
* Karnofsky Performance Status of ≥ 70%.
* Life expectancy of ≥ 3 months.
* Patients must already be taking or begin taking corticosteroids at a stable dose of 4 mg every 6 hours for at least 72 hours prior to catheter placement.
* Patients must be capable of taking, or already taking, anticonvulsant medication.
* Patients must have read, signed, and dated an informed consent according to ICH-GCP, the local regulatory requirement and the rules followed at each institution.

Exclusion Criteria:

Patients fulfilling any of the following criteria should not be enrolled in the study:

* Previous myelosuppressive chemotherapy within the past 4 weeks of the start of the infusion. Patients who have received more than two chemotherapy regimens (single therapy or combination therapy) are ineligible.
* Any form of brain radiation within 10 weeks of the start of the infusion.
* Previous gamma knife radiosurgery, stereotactic radiosurgery, and/or internal radiotherapy, unless the recurrence/progression is histologically confirmed (fine-needle biopsy).
* Prior intracavitary biologic response modifiers or monoclonal antibodies.
* Uncontrolled seizures.
* Bilateral or multifocal tumors.
* Evidence of cerebral uncal herniation.
* Midline brain shift on MRI scan of > 0.5 cm prior to resection; patients with subfalcine herniation may be enrolled.
* Tumors involving the brainstem or cerebellum.
* Diffuse subependymal or CSF disease.
* Women who are pregnant or breast feeding. All women of child-bearing potential should be excluded unless they have a negative pregnancy test and are using adequate contraceptive measures or are surgically sterile. Post-menopausal women must be amenorrheic for at least 12 months to be considered non-childbearing.
* Fertile males not practicing adequate contraception and whose female partners are not using adequate contraceptive protection.
* Prior or concurrent investigational treatment within 30 days of study entry.
* Active infection requiring treatment or having an unexplained febrile illness.
* Systemic diseases or other conditions which may be associated with unacceptable anesthetic/operative risk and/or which would not allow safe completion of this study protocol.
* Prior or concurrent malignancy (curatively treated carcinoma-in-situ or basal cell carcinoma or patients who have been disease free for at least 5 years are eligible).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 56 (Estimated)
Dates: Start 2004-12; Primary Completion 2007-04 (Actual); Study Completion 2007-06 (Actual)

PRIMARY OUTCOMES:
Evaluate TP-38 at a 100 nanograms/mL concentration for sufficient activity | 26 weeks

SECONDARY OUTCOMES:
Efficacy parameters including time to progression, safety, and survival | 26 weeks